CLINICAL TRIAL: NCT06287242
Title: Effectiveness of Matched or Unmatched Cervical and Thoracic Manipulations on Neck Pain: A Randomized Clinical Trial Involving the CTDT (The EMU Manipulation Study)
Brief Title: Validation of the Cervicothoracic Differentiation Test
Acronym: EMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Principal Investigator, Brian Swanson, Principle investigator, associate professor, University of Hartford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-01-282
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain
Keywords: neck pain, manipulation
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded research assistants will perform all baseline and follow-up measures. Investigator providing manipulation is blinded to group allocation (matched/unmatched) Participants will not be told if the CTDT indicates that they would benefit from cervical or thoracic manipulation, and the investigator performing the CTDT will only indicate which region is to be manipulated. All investigators are blinded to the work of the others and submit their results to an additional research assistant who will enter the data in a spreadsheet not accessible to the remainder of the research team until the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- matched manipulation (Active Comparator): For the matched manipulation group, participants with the source of neck pain at the cervical spine determined by the CTDT will receive a cervical manipulation, and participants with the source of neck pain at the thoracic spine determined by the CTDT will receive a thoracic manipulation. The manipulation will be given to the participant's most provocative spinal level as determined by the examiner and side determined by the CTDT. The investigator will be limited to 2 manipulation attempts even if cavitation was not achieved.
  Interventions: Other: spinal manipulation
- unmatched manipulation (Active Comparator): For the unmatched manipulation group, participants with the source of neck pain at the cervical spine determined by the CTDT will receive a thoracic manipulation, and participants with the source of neck pain at the thoracic spine found during the CTDT will receive a cervical manipulation. The manipulation will be given to the most hypomobile spinal level determined by the physical therapist and to the most provocative side found during the CTDT. The investigator will be limited to 2 manipulation attempts even if cavitation was not achieved.
  Interventions: Other: spinal manipulation

INTERVENTIONS:
Other: spinal manipulation — High velocity, low amplitude (HVLA) manipulation of the cervical or thoracic spine

SUMMARY:
The goal of this clinical trial is to compare the effects of two spinal manipulations in adults between the ages of 18-65 based on the results of a non-invasive clinical test. The main question it aims to answer is: • Does matched or unmatched region of manipulation based on the CTDT result in greater reduction of pain levels and improvement in range of motion in adults with neck pain compared to unmatched manipulations? Participants will be asked to:

* rate their pain with neck movement, complete brief questionnaires about their pain,
* have their neck range of motion measured,
* perform a test known as the cervico-thoracic differentiation test (CTDT),
* receive either a cervical or thoracic manipulation,
* repeat the range of motion measurements.
* A second session will occur 7-10 days later where questionnaires and range of motion measures will be repeated.

Researchers will compare the effects of manipulation matched to CTDT test result to individuals in the unmatched CTDT manipulation group to see if the CTDT may indicate which region will provide a greater treatment effect for individuals with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65,
* must report neck pain with a Visual Analogue Scale (VAS) greater than or equal to 3/10.

Exclusion Criteria:

* History of motor vehicle accident (MVA) within the past 6 months,
* hypertension greater than or equal to 160/100,
* non-mechanical neck pain (pain that is not reproducible with movement),
* any past or present history of cancer,
* upper motor neuron (CNS) lesion symptoms ( a positive Clonus sign, Babinski sign, or hyperreflexia of DTR's),
* any infection that originates from the spine
* Current confirmed or suspected pregnancy, or recent postpartum (6 mos),
* known osteoporosis,
* rheumatoid arthritis,
* long-term use of corticosteroids (>6mos),
* history of neck surgery,
* history of vertebral or rib fractures,
* blood clotting disorders,
* connective tissue disorders,
* radicular/neural pain/symptoms. Radicular pain and symptoms would include dermatomal changes (sensory loss or hypersensitization), myotomal changes (weaknesses of muscular along nerve distributions), decreased reflexes (hyporeflexia), pain that travels down the upper extremities, and pain that is referred into the upper extremities.
* clinical signs of instability of the vertebral segments in their neck

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
pain with motion | immediate post intervention, 7-10 days
  pain occurring with the participants most provocative cervical motion as measured on a 100mm visual analog scale (VAS)

SECONDARY OUTCOMES:
pain at rest | immediate post intervention, 7-10 days
  pain occurring with participant at rest
range of motion | immediate post intervention, 7-10 days
  cervical range of motion as measured with the cervical range of motion device (CROM)
neck disability index | 7-10 days post intervention
  questionnaire assessing disability due to neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Brian Swanson, PT, DSc, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No